CLINICAL TRIAL: NCT07076745
Title: Comparative Assessment of High Sensitive CRP and Carotid Stiffness Between Patients With and Without Coronary Slow Flow
Brief Title: High-Sensitive CRP and Carotid Stiffness Between Patients With and Without Coronary Slow Flow
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Remon Saleh Adly, Lecturer of Cardiovascular, Faculty of Medicine, Sohag University, Sohag, Egypt., Sohag University
Other Study IDs: Soh-Med-25-5-6PD
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: High-sensitivity C-reactive Protein; Carotid Stiffness; Coronary Slow Flow

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients diagnosed with coronary slow flow based on corrected thrombolysis in myocardial infarction (TIMI) frame count (cTFC) >27.
  Interventions: Diagnostic Test: High-sensitivity C-reactive protein; Other: Stiffness Measurement
- Control group: Patients with normal coronary angiographic flow and no obstructive coronary artery disease.
  Interventions: Diagnostic Test: High-sensitivity C-reactive protein; Other: Stiffness Measurement

INTERVENTIONS:
Diagnostic Test: High-sensitivity C-reactive protein — High-sensitivity C-reactive protein will be done.
Other: Stiffness Measurement — Measurements will include carotid intima-media thickness (CIMT), systolic (Ds) and diastolic (Dd) diameters, and calculation of stiffness indices:
  * β-stiffness index.
  * Peterson's elastic modulus (Ep).
  * Distensibility coefficient (DC).
  * Compliance coefficient (CC).
  * Strain.

SUMMARY:
This study aims to compare the levels of high-sensitivity C-reactive protein (hs-CRP) and carotid artery stiffness between patients with coronary slow flow phenomenon (CSFP) and those with normal coronary flow.

DETAILED DESCRIPTION:
The coronary slow flow phenomenon (CSFP) is characterized by delayed opacification of the coronary arteries during angiography in the absence of significant epicardial coronary artery disease.

Hypothesis: High-sensitivity C-reactive protein (hs-CRP) is a well-established biomarker of systemic inflammation and has been associated with various cardiovascular conditions. Elevated hs-CRP levels have been observed in patients with CSFP, suggesting an inflammatory component in its pathogenesis. This marker not only predicts future cardiovascular events but may also reflect ongoing vascular inflammation in patients with angiographically normal coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* Patients undergo coronary angiography for evaluation of chest pain or suspected ischemia.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* History of cardiovascular events such as myocardial infarction or stroke.
* Diagnosed autoimmune disorders, chronic hepatic or renal diseases.
* Current or recent infections.
* History of malignancy.
* Patients taking medications known to affect inflammatory markers (e.g., corticosteroids or immunosuppressants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This case-control study will be conducted at Sohag University Hospitals after approval from the institutional ethical committee
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
High Sensitive C-reactive protein | 24 hours post-angiography
  High Sensitive C-reactive protein will be measured.

SECONDARY OUTCOMES:
Stiffness indices | 24 hours post-angiography
  Stiffness indices will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.